CLINICAL TRIAL: NCT05606133
Title: Implementation of Circulating HPV DNA for the Screening and Surveillance of HPV-related Gynecologic Cancers
Brief Title: Circulating Human Papilloma Virus (HPV) DNA for the Screening and Surveillance of Gynecologic Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Naveris (Unknown)
Responsible Party: Principal Investigator, Elena Pereira, Assistant Professor, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-0247
Record Dates: First submitted 2022-08-10; First posted 2022-11-04 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Cervical Dysplasia; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Circulating HPV DNA (Experimental)
  Interventions: Diagnostic Test: NavDx(R)

INTERVENTIONS:
Diagnostic Test: NavDx(R) — NavDx® is a blood test that utilizes digital droplet PCR in order to quantify fragments of tumor-specific DNA shed by HPV-associated cancer cells in the blood. The technology has the ability to distinguish tumor-tissue modified virus particles present in the plasma cell-free DNA from non-cancer associated sources of HPV DNA.

SUMMARY:
Human papilloma virus-related gynecologic malignancies affect over 20,000 women in the United States, and over half a million women globally each year. In addition, approximately 200,000 women are diagnosed with high-grade cervical dysplasia, a pre-cancerous tumor. There is no currently available serum biomarker for these tumors, and surveillance and diagnosis in these patients often requires invasive testing and procedures. The ability to diagnose and monitor for these cancers with a simple blood draw would have a significant impact both here in the US and abroad.

In order to detect circulating tumor-specific HPV DNA, the investigators will collaborate with the molecular diagnostics company, Naveris. Naveris has designed a blood test that utilizes digital droplet polymerase chain reactions (PCR) in order to quantify fragments of tumor-specific DNA that the investigators believe is shed by HPV-associated cancer cells in the blood.

In this pilot study, the investigators will first test whether the quantification of plasma cell-free HPV DNA can distinguish pre-invasive from invasive cervical cancers.

ELIGIBILITY:
Inclusion Criteria:

All patients above age 18, with biopsy proven HPV-related high-grade cervical dysplasia or invasive cervical cancer will be included.

Exclusion Criteria:

Persons who do not meet the above inclusion criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2026-08-10 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
Pre-Treatment Circulating HPV DNA | Week 0
  The presence or absence of ct-HPV DNA
On-Treatment Circulating HPV DNA | Up to 8 weeks
  The presence or absence of ct-HPV DNA
Post-Treatment Circulating HPV DNA | 8-12 weeks
  The presence or absence of ct-HPV DNA

CONTACTS AND LOCATIONS:
Locations (1):
- Lenox Hill Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pereira E, Camacho-Vanegas O, Anand S, Sebra R, Catalina Camacho S, Garnar-Wortzel L, Nair N, Moshier E, Wooten M, Uzilov A, Chen R, Prasad-Hayes M, Zakashansky K, Beddoe AM, Schadt E, Dottino P, Martignetti JA. Personalized Circulating Tumor DNA Biomarkers Dynamically Predict Treatment Response and Survival In Gynecologic Cancers. PLoS One. 2015 Dec 30;10(12):e0145754. doi: 10.1371/journal.pone.0145754. eCollection 2015. PMID 26717006
- [Background] Oh J, Lee HJ, Lee TS, Kim JH, Koh SB, Choi YS. Clinical value of routine serum squamous cell carcinoma antigen in follow-up of patients with locally advanced cervical cancer treated with radiation or chemoradiation. Obstet Gynecol Sci. 2016 Jul;59(4):269-78. doi: 10.5468/ogs.2016.59.4.269. Epub 2016 Jul 13. PMID 27462593
- [Background] Chera BS, Kumar S, Beaty BT, Marron D, Jefferys S, Green R, Goldman EC, Amdur R, Sheets N, Dagan R, Hayes DN, Weiss J, Grilley-Olson JE, Zanation A, Hackman T, Blumberg JM, Patel S, Weissler M, Tan XM, Parker JS, Mendenhall W, Gupta GP. Rapid Clearance Profile of Plasma Circulating Tumor HPV Type 16 DNA during Chemoradiotherapy Correlates with Disease Control in HPV-Associated Oropharyngeal Cancer. Clin Cancer Res. 2019 Aug 1;25(15):4682-4690. doi: 10.1158/1078-0432.CCR-19-0211. Epub 2019 May 14. PMID 31088830
- [Background] Kang Z, Stevanovic S, Hinrichs CS, Cao L. Circulating Cell-free DNA for Metastatic Cervical Cancer Detection, Genotyping, and Monitoring. Clin Cancer Res. 2017 Nov 15;23(22):6856-6862. doi: 10.1158/1078-0432.CCR-17-1553. Epub 2017 Sep 12. PMID 28899967
- [Background] Jeannot E, Becette V, Campitelli M, Calmejane MA, Lappartient E, Ruff E, Saada S, Holmes A, Bellet D, Sastre-Garau X. Circulating human papillomavirus DNA detected using droplet digital PCR in the serum of patients diagnosed with early stage human papillomavirus-associated invasive carcinoma. J Pathol Clin Res. 2016 Jun 28;2(4):201-209. doi: 10.1002/cjp2.47. eCollection 2016 Oct. PMID 27917295
- [Background] Chera BS, Kumar S, Shen C, Amdur R, Dagan R, Green R, Goldman E, Weiss J, Grilley-Olson J, Patel S, Zanation A, Hackman T, Blumberg J, Patel S, Thorp B, Weissler M, Yarbrough W, Sheets N, Mendenhall W, Tan XM, Gupta GP. Plasma Circulating Tumor HPV DNA for the Surveillance of Cancer Recurrence in HPV-Associated Oropharyngeal Cancer. J Clin Oncol. 2020 Apr 1;38(10):1050-1058. doi: 10.1200/JCO.19.02444. Epub 2020 Feb 4. PMID 32017652